CLINICAL TRIAL: NCT03868618
Title: A Multicenter Study to Assess the Safety and Effectiveness of the Genio Dual-sided Hypoglossal Nerve Stimulation System for the Treatment of Obstructive Sleep Apnea in Adults Subjects
Brief Title: Dual-sided Hypoglossal neRvE stimulAtion for the treatMent of Obstructive Sleep Apnea (DREAM)
Acronym: DREAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nyxoah S.A. (Industry)
Collaborators: Nyxoah Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-GEN-002033
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Hypoglossal nerve stimulation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Genio Therapy (Experimental): The Genio™ system is an implantable neurostimulation system comprised of one implanted device
  Interventions: Device: Genio™ system

INTERVENTIONS:
Device: Genio™ system — The Genio™ device is a permanent implant. It is implanted in the chin area and delivers stimulation to both hypoglossal nerve branches (i.e., the left and right branches). The implant does not include a battery or an embedded software and is externally powered.

SUMMARY:
A multicenter study to assess the safety and effectiveness of the Genio dual-sided hypoglossal nerve stimulation system for the treatment of obstructive sleep apnea in adults subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 22 to 75 years (inclusive). Participant cannot be under guardianship, under curatorship or under judicial protection.
2. Body mass index (BMI) ≤ 32 kg/m2.
3. Cricomental space positive (≥ 0 cm). The cricomental space is the distance between the neck and the bisection of a line from the chin to the cricoid membrane when the head is in a neutral position.
4. Has either not tolerated, has failed or refused positive airway pressure (PAP) treatment
5. Moderate to severe OSA (15≤AHI4≤65 where combined central and mixed AHI < 25% of the total AHI) based on a screening PSG.
6. Non-supine AHI > 10 events on the screening PSG or participant has either not tolerated, has failed or refused positional therapy.
7. Written informed consent obtained from the participant prior to performing any study specific procedure.
8. Willing and capable to comply with all study requirements, including specific lifestyle considerations, performing all follow-up visits and sleep studies, evaluation procedures and questionnaires for the whole duration of the trial.
9. Willing to consent to long term follow-up of 5 years post-surgery.

Exclusion Criteria:

1. Inadequately treated sleep disorders other than OSA that would confound functional sleep assessment:

   1. Severe chronic insomnia
   2. Insufficient sleep syndrome (<6 hours sleep per night)
   3. Narcolepsy
   4. Restless legs syndrome
   5. REM behavior disorder
   6. Others deemed sufficient disorders that would confound functional sleep assessment in the judgment of the investigator
2. Night shift worker defined as individual working between the hours of 10:00 pm and 7:00 am at least 3 nights per working week.
3. Taking medications that in the opinion of the investigator may alter consciousness, the pattern of respiration, or sleep architecture.
4. Major anatomical or functional abnormalities that would impair the ability of the Genio System to treat OSA:

   1. Craniofacial abnormalities narrowing the airway or the implantation site
   2. Palatine tonsil size 3+ or 4+ by the Brodsky Classification
   3. Fixed upper airway obstructions (tumor, polyps, nasal obstruction)
   4. Congenital malformations in the airway
   5. Hypoglossal nerve palsy (bilateral limited tongue movement, or unilateral unintended tongue deviation during protrusion)
   6. Existing swallowing difficulty as measured by a score of ≥3 on the EAT-10 questionnaire
   7. Others deemed sufficient to impair the ability of the Genio® System to treat OSA in the judgment of the investigator
5. Significant comorbidities that contraindicate surgery or general anesthesia:

   1. Revised Cardiac Risk Index Class III or IV
   2. Persistent uncontrolled hypertension (defined as systolic pressure 160 mm Hg or a diastolic pressure of 120 mm Hg) despite medications
   3. Coagulopathy or required anticoagulant medications (such as warfarin, clopidogrel (Plavix) or similar; prophylactic aspirin not exclusionary) that cannot be safely stopped in the perioperative period
   4. Degenerative neurological disorder (i.e., Parkinson's disease, Alzheimer's disease)
   5. Acute illness or infection
   6. Diagnosed psychiatric disease (e.g., psychotic illness, uncontrolled major depression or acute anxiety attacks) that prevents participant compliance with the requirements of the investigational study testing
   7. Substance or alcohol abuse history within the previous 3 years. Alcohol and substance abuse are defined as follows:

   i. Alcohol: no days with less than 3 or 4 standard drinks for women and men, respectively

   ii. Substance: the use of any substance in an amount unapproved by the investigator or considered illegal. The drugs most commonly abused include cocaine, marijuana, heroin (or substitution treatment), prescription drugs (especially painkillers), methamphetamines, and various other illegal substances.

   h) Life expectancy less than the primary endpoint study period (12 months post-surgery)

   i) Any other chronic medical illness or condition that contraindicates a surgical procedure or general anesthesia in the judgment of the investigator.
6. Prior surgery or treatments that could compromise the effectiveness of the Genio System:

   1. Airway cancer surgery or radiation
   2. Mandible or maxilla surgery in the previous 5 years (not counting dental treatments)
   3. Other upper airway surgery to remove obstructions related to OSA in the previous 3 months (e.g., uvulopalatopharyngoplasty (UPPP), tonsillectomy, nasal airway surgery)
   4. Prior hypoglossal nerve stimulation device implantation
7. Has an Active Implantable Medical Device (AIMD) even if the device can be temporarily turned off.
8. Participation in another clinical study with an active treatment arm that could confound the results of the DREAM study.
9. Plan to become pregnant, currently pregnant, or breastfeeding during the study period.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in Apnea Hypopnea Index (AHI4%) | 12 months
  percentage of responders at 12 months based on AHI4
Change in Oxyhemoglobin Desaturation Index (ODI4%) | 12 months
  percentage of responders at 12 months based on ODI4

SECONDARY OUTCOMES:
FOSQ-10 | 12 months
  Mean change from baseline to the 12-month visit in FOSQ-10
SNORE-25 | 12 months
  Mean change from baseline to the 12-month visit in SNORE-25
ESS | 12 months
  Mean change from baseline to the 12-month visit in ESS
ODI4 | 12 months
  Mean change from baseline to the 12-month visit in ODI4
SaO2 < 90% | 12 months
  Mean change from baseline to the 12-month visit in SaO2 <90%
AHI4 | 12 months
  Mean change from baseline to the 12-month visit in AHI4

OTHER OUTCOMES:
Safety Objectives | Observed during the study for a period of 12 months post-implantation.
  Incidence of participants with device-related SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Tucker Woodson, MD, Principal Investigator — Medical College of Wisconsin
Locations (21):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - ENT and Allegy Associates South Florida, Boca Raton, Florida
  - University of South Florida-Tampa General Medical Center, Tampa, Florida
  - Advanced Ear Nose & Throat Associates, Atlanta, Georgia
  - CENTA (Center for ENT & Allergy), Carmel, Indiana
  - University of Iowa- Institute for Clinical & Translational Science, Iowa City, Iowa
  - Harvard/ Massachusetts Eye & Ear, Boston, Massachusetts
  - Weill Cornell Medicine Otolaryngology - Head and Neck Surgery, New York, New York
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Thomas Jefferson University Department of Otolaryngology, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Tennessee Health Science Center- Dept. of Otolaryngology, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Wollongong Private Hospital, Wollongong, New South Wales
  - Institute Breathing and Sleep Austin Hospital, Heidelberg, Victoria
  - Hollywood Hospital, Nedlands, Western Australia
- Universitair Ziekenhuis Antwerpen, Antwerp, Belgium
- Technische Universität München, München, Germany

REFERENCES:
- [Derived] Woodson BT, Kent DT, Huntley C, Hancock MK, Van Daele DJ, Boon MS, Huntley TC, Mickelson S, Gillespie MB, Suurna MV, Kacker A, Roy A, MacKay S, Withrow KP, Dedhia RC, Huyett P, Heiser C, Nicola SD, Makori F, Vanderveken OM, Padyha TA, Magalang UJ, Chio E, Kezirian EJ, Lewis R. Bilateral hypoglossal nerve stimulation for obstructive sleep apnea: a nonrandomized clinical trial. J Clin Sleep Med. 2025 Nov 1;21(11):1883-1891. doi: 10.5664/jcsm.11822. PMID 40702817
- [Derived] Woodson BT, Suurna MV, Gillespie MB, Huntley TC, Hancock M, Santos A, Subbaroyan J, Makori F, Fesneau G, Heiser C, Kent DT. Multicentre study conducted across centres in the USA, Europe and Australia to assess the safety and effectiveness of a bilateral hypoglossal nerve stimulation system for the treatment of obstructive sleep apnoea in adults: a protocol for a pivotal, multicentre, open-label, single-arm study. BMJ Open. 2024 Dec 20;14(12):e085218. doi: 10.1136/bmjopen-2024-085218. PMID 39806685